CLINICAL TRIAL: NCT05942365
Title: A Phase 1, Open-Label, Two-Period，Drug Interaction Study Assess the Effects of ZSP1273 Tablets on the Pharmacokinetics of Warfarin and Midazolam
Brief Title: A Drug Interaction Study Assess the Effects of ZSP1273 Tablets on the Pharmacokinetics of Warfarin and Midazolam
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Guangdong Raynovent Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ZSP1273-23-11
Record Dates: First submitted 2023-06-27; First posted 2023-07-12 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Drug Drug Interaction; Warfarin; Midazolam
MeSH Terms: interventions — ZSP1273

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The DDI of ZSP1273 ,Warfarin and Midazolam (Experimental): Warfarin and midazolam will be co-administered alone and in combination with ZSP1273.
  Interventions: Drug: ZSP1273

INTERVENTIONS:
Drug: ZSP1273 — Drug Warfarin oral Drug midazolam oral

SUMMARY:
This study is a single-center, open label phase I clinical study to characterize the DDIs potential of ZSP1273 With Warfarin and Midazolam in Chinese healthy participants. This study also aims to evaluate the safety and tolerability of ZSP1273 in the presence of Warfarin and Midazolam.

ELIGIBILITY:
Inclusion Criteria:

1. Adult, male and female participants, 18 to 55 years of age, inclusive, at first Check-In Visit;
2. Body mass index (BMI) ≥19 to ≤26kg/m2 and total body weight >50 kg(male) or >45kg(female) at Screening (calculated as a function of measured height and weight according to the formula, BMI = kg / m2 where m2 is height in meters squared);
3. Ability to understand and willingness to sign a written informed consent form;
4. Normal physical examination, vital signs, 12-lead ECG, Chest X-ray images (anteroposterior) and clinical laboratory values, or any abnormality that is non-clinically significant.

Exclusion Criteria:

1. Participants with a history of hypersensitivity to study drug(ZSP1273,warfarin, midazolam) or any component of study medication;
2. Participants with a history of and/or signs and symptoms of current abnormal hemostasis or blood dyscrasia or abnormal prothrombin time (PT), international normalized ratio (INR), or activated partial thromboplastin time at screening;
3. Smoking more than 5 cigarettes per day within 3 months prior to screening，or who cannot stop using any tobacco products during the study period;
4. Participants who donated blood/bleeding profusely (> 400 mL) 3 months prior to randomization;
5. Those with clinically significant ECG abnormalities, or QTcF > 450ms in men and QTcF > 470ms in women;
6. Participants who test positive at screening for human immunodeficiency virus (HIV), Hepatitis B surface antigen (HBsAg), Hepatitis C virus (HCV) antibody or Syphilis spirochete-specific antibodies (TPPA);
7. Participants who test positive at Screening and/or admission (Day -1) for alcohol abuse.
8. Females who are pregnant, lactating, or likely to become pregnant during the study.
9. History of dysphagia or any gastrointestinal disorder that affect absorption

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2023-06-25 (Actual); Primary Completion 2023-07-21 (Actual); Study Completion 2023-08-04 (Actual)

PRIMARY OUTCOMES:
S-warfarin Maximum Plasma Concentration [Cmax] | Day1 to Day28
  To assess the effect of steady-state ZSP1273 on the pharmacokinetic (PK) of a single dose of S-warfarin
Midazolam Maximum Plasma Concentration [Cmax] | Day1 to Day28
  To assess the effect of steady-state ZSP1273 on the pharmacokinetic (PK) of a single dose of midazolam and its active metabolite alpha-hydroxymidazolam
S-warfarin Area under the curve[AUC0-inf] | Day1 to Day28
  To assess the effect of steady-state ZSP1273 on the pharmacokinetic (PK) of a single dose of S-warfarin
Midazolam Area under the curve[AUC0-inf] | Day1 to Day28
  To assess the effect of steady-state ZSP1273 on the pharmacokinetic (PK) of a single dose of midazolam and its active metabolite alpha-hydroxymidazolam

SECONDARY OUTCOMES:
Number of participants with adverse events and serious adverse events | Day1 to Day28
  To assess the safety and tolerability of ZSP1273 following single and multiple-dose administration with and without midazolamin+S-warfarin in healthy participates

CONTACTS AND LOCATIONS:
Locations (1):
- the Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, China